CLINICAL TRIAL: NCT02599246
Title: Measured FiO2 With Nasal Canula O2 Versus Noninvasive Ventilation (NIV) With the Same O2 Flow, in COPD Patients the NIV LEAKS Study
Brief Title: FiO2 in Chronic Obstructive Pulmonary Disease (COPD) Patient Normobaric O2 Versus NIV
Acronym: NIVLEAKS
Status: Completed | Type: Observational
Sponsor: Breas Medical S.A.R.L. (Industry)
Responsible Party: Sponsor
Other Study IDs: NIVLEAKS1
Record Dates: First submitted 2015-11-02; First posted 2015-11-06 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2017-01

CONDITIONS: COPD; Home Care; Oxygen Therapy
Keywords: Home ventilator; FiO2; O2; NIV; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to compare pharyngeal FiO2 in day time with nasal normobaric O2 with inhaled FiO2 in the night time with home care ventilator NIV at the same O2 flow.

DETAILED DESCRIPTION:
in a prospective observational study the investigators will register FiO2 in 15 voluntaries COPD patients as following:

* Pharyngeal FiO2 (G5® Philips™ side stream FiO2) with O2 supply through nasal cannula at basal flow (flow needed by patient). In order to compare FiO2s the investigators will measure FiO2 with 150%, 75%, 50% and 25 % of basal Flow
* And FiO2 during nocturnal NIV (pressure support ventilation; Vivo 50®, Bréas™), using facial or nasal masque (Confort Gel® Respironics™). O2 flow will be basal flow.

ELIGIBILITY:
Inclusion Criteria:

* informed consent

Exclusion Criteria:

* acute on chronic respiratory distress

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with chronic obstructive pulmonary disease. With day time oxygenotherapy and nocturnal NIV and O2 supply
Sampling Method: Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2015-11-17 (Actual); Primary Completion 2016-02-22 (Actual); Study Completion 2016-02-24 (Actual)

PRIMARY OUTCOMES:
Difference in FiO2 measured during NIV compared to the FiO2 measured during day time with nasal canula at similar O2 flow | 18 hours

SECONDARY OUTCOMES:
Time spent below different O2 levels during NIV despite constant O2 flow and their correlation to day time FiO2 with nasal canula | 18 hours
levels of O2 adjustment needed to keep FiO2 stable with NIV | 1 hour

CONTACTS AND LOCATIONS:
Overall Officials: Philippe GOUTORBE, MD, Principal Investigator — Military teaching hospital Ste ANNE
Locations (1):
- Military teaching hospital Ste Anne, Toulon, VAR, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Cardinale M, Cungi PJ, Esnault P, Castagna O, Nguyen C, Daranda E, Bordes J, Arnal JM, Meaudre E, Goutorbe P. In COPD, Nocturnal Noninvasive Ventilation Reduces the FIO2 Delivered Compared With Long-Term Oxygen Therapy at the Same Flow. Respir Care. 2020 Dec;65(12):1897-1903. doi: 10.4187/respcare.07570. Epub 2020 Jul 21. PMID 32694183